CLINICAL TRIAL: NCT04894461
Title: Efficacy of Moxibustion in Diabetes Peripheral Neuropathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xiamen University (Other)
Responsible Party: Principal Investigator, Kim Yun Jin, Associate Professor, Xiamen University Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: XiamenU
Record Dates: First submitted 2021-05-16; First posted 2021-05-20 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Peripheral Neuropathy; Diabetic Neuropathies
Keywords: Moxibustion; Peripheral Neuropathy
MeSH Terms: conditions — Peripheral Nervous System Diseases; Diabetic Neuropathies | interventions — Moxibustion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moxibustion (Experimental): Moxibustion treatment sessions eight weeks from the baseline.
  Interventions: Device: Moxibustion
- Waiting (No Intervention): A waiting period of eight weeks by moxibustion treatment sessions in the same way with moxibustion group.

INTERVENTIONS:
Device: Moxibustion — The moxibustion treatment sessions are three times per week for eight weeks. Indirect moxa stick will be used.
  Other Names: Moxa stick
  Arms: Moxibustion

SUMMARY:
This pragmatic randomized controlled study aimed to evaluate the effectiveness and safety of moxibustion therapy on diabetes peripheral neuropathy.

DETAILED DESCRIPTION:
Background: The purpose of this study is to investigate the clinical effects of moxibustion for treating diabetes peripheral neuropathy.

Hypothesis: Subjects who have participated in the moxibustion treatment will have greater improvement in people with diabetes with signs and symptoms of peripheral neuropathy than the control group after 8 weeks.

Design and subjects: A pilot randomized controlled trial. Subjects with diabetes peripheral neuropathy will be recruited from the community. 30 subjects will be randomized to moxibustion groups and control groups in a 1:1 ratio.

Interventions: Subjects in the moxibustion group will receive three times per week for 12 weeks; control groups will be allocated to the waitlist will receive no moxibustion treatments throughout the 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* All patients between 18 and 75 years with diagnosed diabetes mellitus, according to WHO criteria.
* Proven peripheral neuropathy.
* Written consent with documentation that all participants received relevant information about this study is given to the patient.
* The participants must be willing and able to meet the planned visit and meet the planned schedule, including participation in the experimental investigations.

Exclusion Criteria:

* Health professionals' assessment makes the patient have medical or surgical diseases unsuitable to participate in the study.
* Pregnancy or breastfeeding for female patients.
* Competitive conditions that can cause peripheral neuropathy.
* Participants involved in the planning or execution of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Pain assessment measured with Algometry | Measured from Baseline pain at 8 weeks
  For determining sensitivity to pain produced by pressure
Pain assessment measured with the Leeds Assessment of Neuropathic Symptoms and Signs (LANSS) pain scale | Measured from Baseline pain at 8 weeks
  The Leeds assessment of neuropathic symptoms and signs (LANSS) Pain Scale is based on analysis of sensory description and bedside examination of sensory dysfunction, and provides immediate information in clinical settings. The possible scores range from 0 to 24, with a score of 12 or greater considered to be suggestive of neuropathic pain
Pain assessment measured with the Visual Analog Scale | Measured from Baseline pain at 8 weeks
  A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. It is often used in epidemiologic and clinical research to measure the intensity or frequency of various symptoms.
Pain assessment measured with the Neuropathy Pain Scale (NPS) | Measured from Baseline pain at 8 weeks
  Scores are based on patient responses to questions about pain intensity. 0 indicates no pain; 10 indicates the most pain imaginable. The NPS is only for use in patients who have already been diagnosed with neuropathic pain.

SECONDARY OUTCOMES:
Evaluation of functional performance capacity with 6 minutes walking test | Measured from Baseline results at 8 weeks
  It is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.
Evaluation of the Foot and Ankle Ability Measure (FAAM). | Measured from Baseline results at 8 weeks
  It is a self-report outcome instrument developed to assess physical function for individuals with foot and ankle related impairments.
Serum HbA1c | Measured from Baseline results at 8 weeks
  It is provides accurate long-term index of average blood glucose level
Serum Albumin levels | Measured from Baseline results at 8 weeks
  It is measures the amount of the protein albumin in human blood

CONTACTS AND LOCATIONS:
Overall Officials: Linchao Qian, BMed, Study Chair — Xiamen University Malaysia; Muhammad Shahzad Aslam, Ph.D, Study Director — Xiamen University Malaysia

REFERENCES:
- [Derived] Tay JS, Kim YJ. Efficacy of moxibustion in diabetes peripheral neuropathy. Medicine (Baltimore). 2021 Dec 10;100(49):e28173. doi: 10.1097/MD.0000000000028173. PMID 34889293